CLINICAL TRIAL: NCT03656146
Title: Food for Thought: A Randomized Trial of Food Insecurity Screening in the Emergency Department
Brief Title: Food for Thought: Food Insecurity Screening in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 17-013696
Record Dates: First submitted 2018-08-28; First posted 2018-09-04 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Hunger; Child Nutrition Disorders
Keywords: social determinants of health; food insecurity; screening; pediatrics
MeSH Terms: conditions — Child Nutrition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tablet Screening (Active Comparator): Food insecurity screening conducted via electronic tablet
  Interventions: Other: Food Insecurity Screening Tablet
- Verbal Screening (Active Comparator): Food insecurity screening conducted via verbal face-to-face interview
  Interventions: Other: Food Insecurity Screening Verbal

INTERVENTIONS:
Other: Food Insecurity Screening Tablet — The intervention is the type of screening modality used to identify food insecurity: verbal face-to-face, or tablet-based screening
  Arms: Tablet Screening
Other: Food Insecurity Screening Verbal — The intervention is the type of screening modality used to identify food insecurity: verbal face-to-face, or tablet-based screening
  Arms: Verbal Screening

SUMMARY:
This study compares food insecurity disclosure rates in face-to-face interviews versus electronic formats, and explores caregiver preferences regarding screening modality and location, in a large, urban pediatric emergency department. Half of the participants were screened for food insecurity verbally, face-to-face by a research assistant, and half of the participants were screened electronically by a tablet.

DETAILED DESCRIPTION:
Children are disproportionately affected by the rise in poverty rates in the United States, and economic hardships can compromise their development, negatively affect their overall health, and adversely affect their abilities to succeed in school and in life. Food insecurity (FI)-the limited or uncertain availability of nutritionally adequate or safe foods- while strongly associated with poverty, is an independent predictor of poor health outcomes for children.

The Emergency Department (ED) of academic medical centers often serves as a point of care entry for impoverished and high-risk families. Although there is a growing interest in the healthcare system's ability to address Social Determinants of Health (SDH), little is known about food insecurity in the pediatric ED. Additionally, there are limited data on how to implement FI screening into practice in a way that maximizes elicitation of social need, while assuring patient and family comfort.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Adult caregiver accompanying pediatric patient in the Children's Hospital of Philadelphia (CHOP) emergency department

Exclusion Criteria:

* Patient (child) in critical condition
* Patient (child) >18 years of age
* Previously enrolled in study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1818 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2017-11-28 (Actual); Study Completion 2018-01-18 (Actual)

PRIMARY OUTCOMES:
Presence of Food Insecurity | 12 months
  Affirmative response to either of the two, validated screening questions for food insecurity. Investigators measured food insecurity using the validated two-question "Hunger Vital Sign" screening tool, with yes/no responses. These two questions are: within the past 12 months "we worried whether our food would run out before we got money to buy more" and "the food we bought just didn't last and we didn't have money to get more."

SECONDARY OUTCOMES:
Preferred Screening Modality | 4 weeks
  Report of screening modality preference: verbal, tablet, or no preference
Comfort level with screening location | 4 weeks
  Report of comfort with screening in the emergency department and in the primary care setting

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No